CLINICAL TRIAL: NCT02148913
Title: A Phase I Study of Melphalan, Bendamustine, and Carfilzomib for Autologous Hematopoietic Stem Cell Transplantation in Patients With Multiple Myeloma
Brief Title: Phase I: Melphalan, Bendamustine and Carfilzomib for Autologous Transplant in Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corewell Health West (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-067
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1: Carfilzomib 15 mg/m2 (Active Comparator): Carfilzomib 15 mg/m2 on days -2, -1, +5, and +6 IV over 10 minutes.
  Interventions: Drug: Cohort 1: Carfilzomib 15 mg/m2
- Cohort 2: Carfilzomib 20 mg/m2 (Active Comparator): Carfilzomib 20 mg/m2 on days -2, -1, +5, and +6 IV over 10 minutes.
  Interventions: Drug: Cohort 2: Carfilzomib 20 mg/m2
- Cohort 2b: Carfilzomib 20 mg/m2 (Active Comparator): Carfilzomib 20 mg/m2 on days -2, -1 and +5 IV over 10 minutes.
  Interventions: Drug: Cohort 2b: Carfilzomib 20 mg/m2
- Cohort 3: Carfilzomib 27mgm2 (Active Comparator): Carfilzomib 27 mg/m2 on days -2, -1 and +5 IV over 10 minutes.
  Interventions: Drug: Cohort 3b: Carfilzomib 27 mg/m2

INTERVENTIONS:
Drug: Cohort 1: Carfilzomib 15 mg/m2 — Carfilzomib 20 mg/m2 on days -29, -28, -22, -21, -15, and -14 Bendamustine 120 mg/m2 on day -2 and 100 mg/m2 day -1 Melphalan 100 mg/m2 on day -2 and day -1 Carfilzomib 15 mg/m2 on day -2, -1, + 5 and +6
  Other Names: Carfilzomib - Kyprolis; Bendamustine - Treanda; Melphalan - Alkeran
  Arms: Cohort 1: Carfilzomib 15 mg/m2
Drug: Cohort 2: Carfilzomib 20 mg/m2 — Carfilzomib 20 mg/m2 on days -29, -28, -22, -21, -15, and -14 Bendamustine 120 mg/m2 on day -2 and 100 mg/m2 day -1 Melphalan 100 mg/m2 on day -2 and day -1 Carfilzomib 20 mg/m2 on day -2, -1, + 5 and +6
  Other Names: Carfilzomib - Kyprolis; Bendamustine - Treanda; Melphalan - Alkeran
  Arms: Cohort 2: Carfilzomib 20 mg/m2
Drug: Cohort 2b: Carfilzomib 20 mg/m2 — Carfilzomib 20 mg/m2 on days -29, -28, -22, -21, -15, and -14 Bendamustine 120 mg/m2 on day -2 and 100 mg/m2 day -1 Melphalan 140 mg/m2 on day -1 Carfilzomib 20 mg/m2 on day -2, -1 and + 5
  Other Names: Carfilzomib - Kyprolis; Bendamustine - Treanda; Melphalan - Alkeran
  Arms: Cohort 2b: Carfilzomib 20 mg/m2
Drug: Cohort 3b: Carfilzomib 27 mg/m2 — Carfilzomib 20 mg/m2 on days -29, -28, -22, -21, -15, and -14 Bendamustine 120 mg/m2 on day -2 and 100 mg/m2 day -1 Melphalan 140 mg/m2 on day -1 Carfilzomib 27 mg/m2 on day -2, -1 and + 5
  Other Names: Carfilzomib - Kyprolis; Bendamustine - Treanda; Melphalan - Alkeran
  Arms: Cohort 3: Carfilzomib 27mgm2

SUMMARY:
This is a phase I clinical trial. Patients with a diagnosis of multiple myeloma undergoing autologous transplantation will receive a preparative regimen of melphalan, bendamustine, and carfilzomib. We hypothesize that the addition of carfilzomib to a conditioning regimen of melphalan and bendamustine in the setting of autologous transplantation for multiple myeloma is feasible and safe.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma
* At least 2 x 106 CD34+ cells/kg have been collected from the patient and cryopreserved for ASCT
* Greater than 18 years
* Karnofsky score greater than 70%
* No evidence of progressive bacterial, viral, or fungal infection
* Absolute neutrophil count above 1000
* Platelet count above 50,000
* Hemoglobin above 8 g/dL
* Creatinine clearance greater than 50 mL/min
* Total bilirubin, ALT, and AST less than 2 x the upper limit of normal
* Alkaline phosphatase less than or equal to 250 IU/L
* Left Ventricular Ejection Fraction (LVEF) greater than or equal to 45%
* Adjusted Carbon Monoxide Diffusing Capacity (DLCO) greater than or equal to 60%
* Negative HIV serology
* Recovered from toxicity of previous chemotherapy (excludes grade 1 neurotoxicity and hematological toxicity)
* Patients with a pre-transplant disease status consistent with a very good partial response (VGPR), partial response (PR), stable disease (SD), progressive disease (PD), or relapse from complete remission (CR).

Exclusion Criteria:

* Patients who are refractory to carfilzomib. Refractory is defined as disease progression while on carfilzomib therapy after receiving at least two cycles of treatment.
* Patients with a complete response (CR) (including near CR and stringent CR) to conventional induction therapy and proceeding to transplantation.
* Pregnant or nursing females or women of reproductive capability who are unwilling to use effective contraception. A woman of reproductive capability is one who has not undergone a hysterectomy (removal of the womb), has not had both ovaries removed, or has not been post-menopausal (stopped menstrual periods) for more than 24 months in a row.
* Male subjects who refuse to practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse. This must be done even if they are surgically sterilized (ie, post-vasectomy).
* Patient with Grade 2 peripheral neuropathy
* Inability to provide informed consent
* Patient had myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
* Known allergies to any of the components of the investigational treatment regimen or required ancillary treatments.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 3 years of enrollment (with the exception of non-melanoma skin cancer).
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muneer H Abidi, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health, Grand Rapids, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted using a standard 3+3 phase I design. If dose-limiting toxicity (DLT) occurred in 1 out of 3 patients, 3 additional patients were enrolled at that same dose level. Dose escalation was permitted if DLT did not occur in more than 0 out of 3, or 1 out of 6 patients
Period: Overall Study
Arm/Group | Cohort 1: Carfilzomib 15 mg/m2 | Cohort 2: Carfilzomib 20 mg/m2 | Cohort 2b: Carfilzomib 20 mg/m2 | Cohort 3: Carfilzomib 27mgm2
Started | 3 | 3 | 3 | 9
Completed | 3 | 2 | 3 | 9
Not Completed | 0 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Carfilzomib 15 mg/m2 | Cohort 2: Carfilzomib 20 mg/m2 | Cohort 2b: Carfilzomib 20 mg/m2 | Cohort 3: Carfilzomib 27mgm2 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 2 | 7 | 14
  >=65 years | 0 | 1 | 1 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 3 | 7
  Male | 1 | 1 | 3 | 6 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Absence of Dose Limiting Toxicity
Description: An absence of neutrophil engraftment by Day +22, absence of platelet engraftment by Day +35, and any grade 4 GI toxicity or any >/= grade 3 non-hematologic toxicity as defined by the common toxicity criteria, which is deemed by the DSMB as probably related to the study protocol.
Time Frame: Assessed daily (while inpatient) through clinical and laboratory examinations up to 90 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Carfilzomib 15 mg/m2 | Cohort 2: Carfilzomib 20 mg/m2 | Cohort 2b: Carfilzomib 20 mg/m2 | Cohort 3: Carfilzomib 27mgm2
Number analyzed (Participants) | 3 | 3 | 3 | 9
Participants | 3 | 1 | 3 | 9

2. Secondary Outcome: Neutrophil Engraftment
Description: Engraftment of Neutrophils: ANC recovery is defined as an absolute neutrophil count (ANC) of ≥ 0.5 x 109/L for three consecutive laboratory values obtained on different days. The day used as neutrophil engraftment is the date of the first of three laboratory values.
  Graft Failure: Graft failure includes failure to achieve neutrophil engraftment by day 22.
Time Frame: Assessed daily (while inpatient) through clinical and laboratory examinations up to 90 days.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort 1: Carfilzomib 15 mg/m2 | Cohort 2: Carfilzomib 20 mg/m2 | Cohort 2b: Carfilzomib 20 mg/m2 | Cohort 3: Carfilzomib 27mgm2
Number analyzed (Participants) | 3 | 3 | 3 | 9
days | 11.33 (0.58) | 12.67 (2.08) | 12 (0) | 12.11 (0.78)

3. Secondary Outcome: Platelet Engraftment
Description: Engraftment of Platelets: Platelet engraftment is defined as a platelet count ≥ 20 x 109/L for 3 consecutive measurements obtained on different days. The patient must not have received a platelet infusion for seven consecutive days prior to the first day being considered. The day used as platelet engraftment is the date of the first of three laboratory values.
Time Frame: Assessed daily (while inpatient) through clinical and laboratory examinations up to 90 days.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cohort 1: Carfilzomib 15 mg/m2 | Cohort 2: Carfilzomib 20 mg/m2 | Cohort 2b: Carfilzomib 20 mg/m2 | Cohort 3: Carfilzomib 27mgm2
Number analyzed (Participants) | 3 | 2 | 3 | 9
days | 17 (2.65) | 15.5 (0.71) | 15.67 (3.51) | 15.89 (1.96)

4. Other Pre Specified Outcome: Response Rate
Description: Find the response rate of the combination of melphalan, bendamustine, and carfilzomib as a conditioning regimen in patients with multiple myeloma undergoing autologous transplantation.
Time Frame: Disease assessment at day +100, +180, and +365 (+/- 7 days).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Carfilzomib 15 mg/m2 | Cohort 2: Carfilzomib 20 mg/m2 | Cohort 2b: Carfilzomib 20 mg/m2 | Cohort 3: Carfilzomib 27mgm2
Number analyzed (Participants) | 3 | 2 | 3 | 9
Participants
  complete response | 1 | 1 | 0 | 2
  very good partial response | 2 | 0 | 1 | 2
  partial response | 0 | 1 | 1 | 2
  progressive disease | 0 | 0 | 1 | 3

ADVERSE EVENTS:
Time Frame: CBC, CMP, BUN, creatinine labs, and LFT were then measured at least weekly until day +100. Daily physical examination, including toxicity assessments were conducted until discharge and then weekly until day +100. Disease assessments were conducted at day +100, +180, and +365 (+/- 7 days).
Description: CTCAE v4.0
Arm/Group | Cohort 1: Carfilzomib 15 mg/m2 | Cohort 2: Carfilzomib 20 mg/m2 | Cohort 2b: Carfilzomib 20 mg/m2 | Cohort 3: Carfilzomib 27mgm2
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 0/3 | 0/9
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Carfilzomib 15 mg/m2 (N=3) | Cohort 2: Carfilzomib 20 mg/m2 (N=3) | Cohort 2b: Carfilzomib 20 mg/m2 (N=3) | Cohort 3: Carfilzomib 27mgm2 (N=9)
Acute Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — developed grade 4 acute respiratory distress, grade 3 prolonged intubation, and grade 3 pneumonia. deteriorated neurologically and subsequently was shown to have experienced a brain hemorrhage and expired on day +44
Septic Shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — developed grade 4 febrile neutropenia, and several grade 3 events secondary to septic shock (grade 3 elevated troponin T, grade 3 hypotension, and grade 3 left ventricular dysfunction) from Escherichia coli enteritis.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Carfilzomib 15 mg/m2 (N=3) | Cohort 2: Carfilzomib 20 mg/m2 (N=3) | Cohort 2b: Carfilzomib 20 mg/m2 (N=3) | Cohort 3: Carfilzomib 27mgm2 (N=9)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 6 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
mucositis/esophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
partial ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hypophosphatemia (Investigations) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
hypocalcemia (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
hypokalemia (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
hypermagnesemia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
elevated ALT (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
elevated AST (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
elevated serum creatinine (Investigations) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
elevated bilirubin (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
elevated alkaline phosphatase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
febrile neutropenia (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 4 (4)
pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
fever of unknown origin (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
typhlitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
elevated troponin T (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
LV systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
arrhythmia--a fib (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
edema (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
decreased EF (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AV block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
prolonged QTc interval (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
prolonged intubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT02148913/Prot_000.pdf